CLINICAL TRIAL: NCT05816447
Title: Patients' Perception of Climate Change and Healthcare - a Cross-section Cohort Study in a Single Institution in Canada
Brief Title: Patients' Perception of Climate Change and Healthcare
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00128836
Record Dates: First submitted 2023-03-31; First posted 2023-04-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Perception, Self
Keywords: Environmental sustainability; Anesthesia; Healthcare
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: interview — Interview patient's perception

SUMMARY:
This study aims to investigate the patients' perception of the negative impact of the healthcare industry on climate change, their attitude of climate change and their health, and their view of seeing a change in the healthcare system to reduce climate change.

DETAILED DESCRIPTION:
Climate change is a threat to human health which in turn increases burden on our healthcare system. Healthcare is also a very polluted industry which has a huge contribution to climate change. It is important to take action and the intergovernmental panel on climate change (IPCC) has put out a warning of 'Code Red for Humanity' urging immediate action from all of humanity to combat climate change. This is important because if no action is taken, irreversible damage might result on our planet which will become a challenge in terms of living conditions, food source, and health.

Therefore, this study aims to investigate the patients' perception of the negative impact of the healthcare industry on climate change, their attitude of climate change and their health, and their view of seeing a change in the healthcare system to reduce climate change. This will produce data on the knowledge gap in our patients and thereby empower them to request and target our education for patients, and in turn encourage the healthcare system to reflect on their environmental sustainable practices.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients > age of 18 years old
* Willing and able to read/listen and understand English, on the hospital ward ie. Not Emergency Department

Exclusion Criteria:

* Patient refusal
* Patients are unable to consent
* Confusion or disorientated in time, space and person

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients at the hospital
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Patients' awareness of climate change from the healthcare industry | Baseline
  If patients are aware (Yes or No) of climate change effects from healthcare industry via a questionnaire

SECONDARY OUTCOMES:
To evaluate their attitude on climate change, view of change in the healthcare system to reduce climate change | Baseline
  To evaluate their attitude on climate change, as well as their view of seeing a change in the healthcare system to reduce climate change. There are a set of interview questions (questionnaires) in a Likert scale or Yes/No to assess this as this is a qualitative study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No